CLINICAL TRIAL: NCT05608564
Title: The Impact of Local vs. Systemic Adjuvant Antibiotics During Non-surgical Periodontitis Therapy on Clinical Parameters, Bacterial Count and Cytokine Levels - a Randomized Clinical Trial
Brief Title: Local and Systemic Antimicrobials in Non-surgical Periodontal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Iva Milinkovic, Assistant Professor, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22.10.1980
Record Dates: First submitted 2022-10-24; First posted 2022-11-08 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Periodontitis
Keywords: local antibiotics; systemic antibiotics
MeSH Terms: conditions — Periodontitis | interventions — Piperacillin; Tazobactam; Amoxicillin; Metronidazole

STUDY DESIGN:
Intervention Model Description: After the non-surgical periodontal treatment, the test group will be treated with local antibiotics, while the control group will be treated with systemic antibiotics. Randomization will be performed using randomization envelopes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local antibiotic group (Experimental): A combination of Piperacillin and Tazobactam in gel form is applied using a syringe and a flexible blunt needle into the periodontal pockets 24 hours after the non-surgical periodontal therapy. After administration, the dry field should be maintained for 5 minutes and the patient should not rinse the oral cavity for 15 minutes.
  Interventions: Procedure: Piperacillin and Tazobactam in gel form
- Systemic antibiotic group (Active Comparator): Amoxicillin (500mg, 3 times a day, 7 days) and Metronidazole (400mg, 3 times a day, 7 days) per os at the beginning of non-surgical treatment.
  Interventions: Procedure: Amoxicillin and Metronidazole

INTERVENTIONS:
Procedure: Piperacillin and Tazobactam in gel form — After non-surgical periodontal treatment, the test group will receive local antibiotics.
  Other Names: Gelcide
  Arms: Local antibiotic group
Procedure: Amoxicillin and Metronidazole — After non-surgical periodontal treatment, the control group will receive systemic antibiotics.
  Other Names: Amoxicillin and Orvagyl
  Arms: Systemic antibiotic group

SUMMARY:
The main treatment of every patient with periodontitis is non-surgical periodontal treatment (NSPT) with the ultimate goal to arrest inflammation. Given the biofilm microorganisms associated etiology of the periodontitis, NSPT can be combined with adjunctive antimicrobial therapy. Hence, this randomized clinical trial aims to compare the clinical and microbiological effectiveness and relative expression levels (REL) of proinflammatory cytokines tumor necrosis factor-alpha (TNF-α) and interleukin-17 (IL-17) between local and systemic antibiotics as adjunctive therapy to NSPT in patents with periodontitis stage 3.

DETAILED DESCRIPTION:
Study protocol:

This randomized clinical study will include 40 patients diagnosed with periodontitis stage 3. The investigation will be conducted at the Department of Periodontology and Oral Medicine, at the School of Dental Medicine, University of Belgrade. The laboratory part of the research will be carried out at the Department of Human genetics, at the School of Dental Medicine, University of Belgrade. Patients will be divided into two groups. The test group will consist of 20 patients who will be prescribed a local antibiotic (LA group), while the control group will consist of 20 patients who will be prescribed systemic antibiotic therapy (SA group). The division of patients into groups will be done with randomization envelopes after the diagnostic procedure.

Upon clinical examination, clinical periodontal parameters such as periodontal probing depth (PPD), clinical attachment level (CAL), bleeding on probing (BOP), and plaque index (PI) will be recorded for each patient around every tooth. Previous to treatment, subgingival crevicular fluid will be sampled with paper points from periodontal pockets for laboratory analysis.

Sampling will be performed as follows: first, a relatively dry working field will be established using paper water rollers and air jets, and then 3 paper points (number 30 - marked in blue) will be applied for 30 seconds in the periodontal pocket area of the selected premolar/molar tooth with a depth of more than 5mm. The procedure will be repeated immediately in the same region, to obtain duplicate samples. After that, the paper points will be placed in Eppendorf tubes and immediately transported to the basic research laboratory, where they will be stored at a temperature of -80 degrees Celsius and where microbiological and molecular analyses will be carried out.

After sampling, all patients will undergo a non-surgical phase of periodontal therapy, following a Full-mouth disinfection protocol. Six months after the NSPT, at the follow-up, clinical examination, detection of clinical parameters, and sampling procedure will be repeated. In the LA group, antibiotics will be applied after the NSPT, while in the SA group therapy will be prescribed at the beginning of the treatment. Locally will be applied a combination of piperacillin and tazobactam in gel form (Gelcide ®, Italmed MedTechDental, Florence, Italy) designed for use in the subgingival region. The local antibiotic will be applied into the periodontal pockets, using a syringe and a flexible blunt needle, 24 hours after the NSPT. The administration will be done by quadrants, following the principles of a dry work field, and after application, the dry field should be maintained for 5 minutes. After this procedure, the patient should not rinse the oral cavity for 15 minutes. For systemic use in the SA group, patients will receive a combination of Amoxicillin (Amoxicillin ®, 500mg, 3 times a day, 7 days) and Metronidazole (Orvagyl ®, 400mg, 3 times a day, 7 days) for oral use.

Total bacterial count (TBC) and REL of proinflammatory cytokines TNF-α and IL-17 will be detected using the quantitative real-time polymerase chain reaction (qPCR) in a basic research laboratory at the Department of Human genetics, at the School of Dental Medicine, University of Belgrade.

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes, 18 - 45 years old
2. Willingness to participate in the research, comply with all the study protocols, and sign an informed consent;
3. Active periodontitis stage II and III according to the criteria of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions;
4. Non-smokers and light smokers (up to 10 cigarettes per day).

Exclusion Criteria:

1. Presence of systemic diseases known to affect the tooth-supporting apparatus and bone metabolism (such as uncontrolled diabetes mellitus, cancer, immunodeficiency, metabolic bone diseases);
2. Patients receiving an immunosuppressive, anti-resorptive, or anti-inflammatory therapy;
3. Allergy to penicillin;
4. Patients who had undergone periodontal therapy within the last 6 months;
5. Use of local and/or systemic antimicrobial agents within the last 6 months;
6. Use of oral anti-plaque mouthwash at least one month prior to the study;
7. Alcohol or drug abuse;
8. Pregnancy or lactation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2024-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iva Z Milinkovic, DDS, PhD, Principal Investigator — School of Dental Medicine, University of Belgrade, Department of Periodontology and Oral Medicine
Locations (1):
- Department of Periodontology, School of Dental Medicine, University of Belgrade, Belgrade, Serbia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 38 participants screened at the Department of Periodontology and Oral Medicine at the School of Dental Medicine University of Belgrade, 38 participants were enrolled
Pre-assignment Details: All 38 participants who met the inclusion criteria were enrolled and directly assigned to study groups without a pre-assignment phase.
Groups:
- Open- Label Local Antibiotic Group: A combination of Piperacillin and Tazobactam in gel form is applied using a syringe and a flexible blunt needle into the periodontal pockets 24 hours after the non-surgical periodontal therapy. After administration, the dry field should be maintained for 5 minutes and the patient should not rinse the oral cavity for 15 minutes.
  Piperacillin and Tazobactam in gel form: After non-surgical periodontal treatment, the test group will receive local antibiotics.
- Open- Label Systemic Antibotic Group: Amoxicillin (500mg, 3 times a day, 7 days) and Metronidazole (400mg, 3 times a day, 7 days) per os at the beginning of non-surgical treatment.
  Amoxicillin and Metronidazole: After non-surgical periodontal treatment, the control group will receive systemic antibiotics.
Period: Overall Study
Arm/Group | Open- Label Local Antibiotic Group | Open- Label Systemic Antibotic Group
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Thirty-eight patients diagnosed with stage III periodontitis were included in the study. They were evenly distributed into two groups: 19 in the LA group and 19 in the SA group. The cohort comprised 23 female and 15 male participants, with an age range of 24 to 40 years.
Groups:
- Systemic Antibotic Group: Amoxicillin (500mg, 3 times a day, 7 days) and Metronidazole (400mg, 3 times a day, 7 days) per os at the beginning of non-surgical treatment.
  Amoxicillin and Metronidazole: After non-surgical periodontal treatment, the control group will receive systemic antibiotics.
- Total: Total of all reporting groups
Arm/Group | Local Antibiotic Group | Systemic Antibotic Group | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Full Range); unit: years] | 33.59 [24 to 40] | 36.06 [27 to 40] | 34.83 [24 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 8 | 7 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Data was collected in specified questioners and entered in the Excel table.
  participants
    Serbia | 19 | 19 | 38
PPD baseline [Mean (Standard Deviation); unit: mm] — PPD was detected with the periodontal probe at 6 sites around each present tooth in millimeters (mm).
  mm | 3.932 (0.5355) | 4.082 (0.5812) | 4.007 (0.556)
CAL baseline [Mean (Standard Deviation); unit: mm] — CAL was detected with the periodontal probe at 6 sites around each present tooth in millimeters (mm).
  mm | 4.4 (0.8452) | 4.494 (0.7677) | 4.447 (0.8088)
BOP baseline [Mean (Standard Deviation); unit: percentage] — BOP was detected with the periodontal probe at 6 sites around each present tooth; it was recorded as present (1) or not (0) at each site, and expressed in percentage (%).
  percentage | 0.6311 (0.1214) | 0.6794 (0.1861) | 0.655 (0.157)
PI baseline [Mean (Standard Deviation); unit: percentage] — PI was detected with the periodontal probe at 6 sites around each present tooth; it was recorded as present (1) or not (0) at each site, and expressed in percentage (%).
  percentage | 0.6537 (0.1283) | 0.7041 (0.2525) | 0.670 (0.119)
TBL [Mean (Standard Deviation); unit: CFU/mL] — Gingival crevicular fluid (GCF) was collected from periodontal pockets using sterile paper strips to analyze the total bacterial load (TBL). TBL was then quantified using real-time polymerase chain reaction (qPCR) and expressed in colony-forming units per milliliter (CFU/mL).
  CFU/mL | 1.87 (5.44) | 1.79 (5.54) | 1.80 (5.42)
TNF-α [Mean (Standard Deviation); unit: ng/mL] — Gingival crevicular fluid (GCF) was collected from periodontal pockets using sterile paper strips. The relative expression level (REL) of tumor necrosis factor-alpha (TNF-α) was then quantified using real-time polymerase chain reaction (qPCR) and expressed in nanograms per milliliter (ng/mL).
  ng/mL | 0.03347 (0.01475) | 0.05048 (0.06895) | 0.042 (0.050)
IL-17 [Mean (Standard Deviation); unit: ng/mL] — Gingival crevicular fluid (GCF) was collected from periodontal pockets using sterile paper strips. The relative expression level (REL) of interleukin 17 (IL-17) was then quantified using real-time polymerase chain reaction (qPCR) and expressed in nanograms per milliliter (ng/mL).
  ng/mL | 0.008072 (0.004611) | 0.007164 (0.008121) | 0.00762 (0.00653)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pocket Probing Depth (PPD)
Description: Pocket probing depth (PPD) was measured using a periodontal probe at 6 sites per tooth, recorded in millimeters (mm), at baseline and at 6-month follow-up. This measure was used to compare outcomes between local and systemic antimicrobial therapies.
Time Frame: baseline and 6 months follow up
Population: All patients from both groups, at baseline and 6 months recall.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Open- Label Local Antibiotic Group | Open- Label Systemic Antibotic Group
Number analyzed (Participants) | 19 | 19
mm
  PPD baseline | 3.932 (0.5355) | 4.082 (0.5812)
  PPD 6 months | 3.253 (0.5048) | 3.294 (0.5471)

2. Primary Outcome: Change in Clinical Attachment Level (CAL)
Description: as for outcome 1
Time Frame: baseline and 6 months follow up
Population: All patients from both groups, at baseline and 6 months recall.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Open- Label Local Antibiotic Group | Open- Label Systemic Antibotic Group
Number analyzed (Participants) | 19 | 19
mm
  CAL baseline | 4.4 (0.8452) | 4.494 (0.7677)
  CAL 6 months | 3.832 (0.9062) | 4.035 (0.8031)

3. Primary Outcome: Change in Bleeding On Probing (BOP)
Description: Bleeding on probing (BOP) was assessed using a periodontal probe at 6 sites around each present tooth during baseline and 6-month follow-up clinical examinations. BOP was recorded as present (1) or absent (0) at each site, and expressed as a percentage (%).
Time Frame: baseline and 6 months follow up
Population: All patients from both groups, at baseline and 6 months recall.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Open- Label Local Antibiotic Group | Open- Label Systemic Antibotic Group
Number analyzed (Participants) | 19 | 19
percentage
  BOP baseline | 0.6311 (0.1214) | 0.6794 (0.1861)
  BOP 6 months | 0.1232 (0.0844) | 0.6794 (0.1861)

4. Primary Outcome: Change in Plaque Index (PI)
Description: Plaque Index (PI) was assessed using a periodontal probe at 6 sites around each present tooth during baseline and 6-month follow-up clinical examinations. BOP was recorded as present (1) or absent (0) at each site, and expressed as a percentage (%).
Time Frame: baseline and 6 months follow up
Population: All patients from both groups, at baseline and 6 months recall.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Open- Label Local Antibiotic Group | Open- Label Systemic Antibotic Group
Number analyzed (Participants) | 19 | 19
percentage
  PI baseline | 0.6537 (0.1283) | 0.7041 (0.2525)
  PI 6 months | 0.1005 (0.06399) | 0.1147 (0.04048)

5. Secondary Outcome: Changes in Relative Expression Levels of Tumor Necrois Factor Alpha (TNF-α)
Description: Relative expression levels (REL) of TNF-α were assessed in gingival crevicular fluid (GCF) samples collected from periodontal pockets at baseline and 6-month follow-up. GCF was obtained using sterile paper strips, and TNF-α levels were quantified using the real-time polymerase chain reaction (qPCR) method. Results were expressed in nanograms per milliliter (ng/mL) to compare local and systemic antimicrobial therapy groups.
Time Frame: baseline and 6 months follow up
Population: All patients from both groups, at baseline and 6 months recall.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Open- Label Local Antibiotic Group | Open- Label Systemic Antibotic Group
Number analyzed (Participants) | 19 | 19
ng/mL
  TNF-α baseline | 0.03347 (0.01475) | 0.05048 (0.06895)
  TNF-α 6 months | 0.03483 (0.03704) | 0.02407 (0.01503)

6. Secondary Outcome: Change in Total Bacterial Load (TBL)
Description: Total bacterial load (TBL) was assessed in gingival crevicular fluid (GCF) samples collected from periodontal pockets at baseline and at the 6-month follow-up. GCF was obtained using sterile paper strips, and bacterial quantification was performed using the real-time polymerase chain reaction (qPCR) method. Results were expressed in colony-forming units per milliliter (CFU/mL) to evaluate differences between local and systemic antimicrobial therapies.
Time Frame: baseline and 6 months follow up
Population: All patients from both groups, at baseline and 6 months recall.
Measure: Mean (Standard Deviation); unit: CFU/mL
Arm/Group | Open- Label Local Antibiotic Group | Open- Label Systemic Antibotic Group
Number analyzed (Participants) | 19 | 19
CFU/mL
  TBL baseline | 1.87 (5.44) | 1.79 (5.54)
  TBL 6 months | 1.71 (4.27) | 2.00 (4.61)

7. Secondary Outcome: Changes in Relative Expression Levels of IL-17
Description: Relative expression levels (REL) of interleukin-17 (IL-17) were assessed in gingival crevicular fluid (GCF) samples collected from periodontal pockets at baseline and at the 6-month follow-up. GCF was obtained using sterile paper strips, and REL of IL-17 was quantified using the real-time polymerase chain reaction (qPCR) method. Results were expressed in nanograms per milliliter (ng/mL) to compare local and systemic antimicrobial therapies.
Time Frame: baseline and 6 months follow up
Population: All patients from both groups, at baseline and 6 months recall.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Open- Label Local Antibiotic Group | Open- Label Systemic Antibotic Group
Number analyzed (Participants) | 19 | 19
ng/mL
  IL-17 baseline | 0.008072 (0.004611) | 0.007164 (0.008121)
  IL-17 6 months | 0.007358 (0.005917) | 0.00455 (0.00391)

ADVERSE EVENTS:
Time Frame: Data were collected in 6 months follow-up period
Arm/Group | Open- Label Local Antibiotic Group | Open- Label Systemic Antibotic Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT05608564/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT05608564/ICF_001.pdf